CLINICAL TRIAL: NCT07048535
Title: CAR T-cell Long-Term Follow-Up, Quality of Life and Adverse Reactions
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CONQUER
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: B-Cell Acute Lymphoblastic Leukemia (B-ALL)
Keywords: B-Cell Acute Lymphoblastic Leukemia; B-ALL; Survivorship
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine:
  The collected blood and urine samples will be stored according to the clinical and research infrastructure of the institutional tissue bank - SJLIFE. The samples will be tagged accordingly and will be only released to fulfill future objectives of the CONQUER protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To learn more about the long-term health in patients treated for B-Cell Acute Lymphoblastic Leukemia (B-ALL) with Cluster of Differentiation antigen 19 (CD19)

-redirected chimeric antigen receptor (CAR) T-cells.

Primary Objective:

To evaluate the feasibility of conducting standardized clinical assessments of pediatric, adolescent and young adult (AYA) B-ALL survivors post CD19-CAR T-cell therapy, treated at multiple institutions, leveraging the St Jude Lifetime Cohort (SJLIFE) clinical and research infrastructure.

Exploratory Objectives:

* To describe the prevalence of persistent and new/late-onset health conditions developing ≥2-years post CD19-CAR T-cell therapy in survivors of pediatric and AYA B-ALL.
* To characterize neurocognitive and neurologic function in survivors ≥2-years post CD19- CAR T-cell therapy.
* To characterize immune health in survivors ≥2-years post CD19-CAR T-cell therapy.
* To characterize functional status in survivors ≥2-years post CD19-CAR T-cell therapy.

DETAILED DESCRIPTION:
Advances in cancer immunotherapies, including CD19-redirected chimeric antigen receptor (CAR) T-cells, are changing the long-term outcome for B-ALL cancer patients.

The late effects of these treatments have not been investigated and the impact of this therapy on survivors' long-term outcomes and overall well-being is unknown.

The purpose of this study is to determine the feasibility of studying late effects following CAR T-cell therapy through a prospective, observational study for children, adolescent, and young adult (AYA) survivors who are ≥2-years post CD19-CAR T-cell infusion. The study will be the first study of late effects following CAR T-cell therapy recruiting B-ALL survivors from across the United States.

Eligible study participants will participate in a comprehensive health assessment. These assessments will include history and physical examination, laboratory studies, a brain MRI, physical performance testing, and neurocognitive testing. The CONQUER study will focus specific attention on data relevant to CD19-CAR T-cell therapy, including immune function.

ELIGIBILITY:
Inclusion Criteria:

* ≤ 26-years old at the time of the first CAR treatment
* Receipt of a CD19-containing CAR T-cell product (investigational or commercial) for B- ALL
* Receipt of one unique CAR product (reinfusion of same product allowed)
* Sustained remission without subsequent therapy post-CAR (exception= post-CAR consolidative HCT)
* Receipt of only one prior HCT (inclusive of pre- or post-CAR)
* ≥ 2-years post last CAR T-cell infusion

Exclusion Criteria:

* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants who meet eligibility criteria and consent to enrollment on the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the feasibility of conducting standardized clinical assessments of pediatric and AYA B-ALL survivors post CD19-CAR T-cell therapy | Through study completion, approximately 5 years
  Estimation of participation rate

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Talleur, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols